CLINICAL TRIAL: NCT04501042
Title: Investigation on Novel Route of Gut Microbiota Products for Bariatric Surgery to Improve Non-alcoholic Steatohepatitis and Development on Therapeutic Implications
Brief Title: Investigation on the Role of Gut-liver Axis for Non-alcoholic Steatohepatitis Through Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201903037RIND
Record Dates: First submitted 2020-07-22; First posted 2020-08-06 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2021-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; Bariatric Surgery
Keywords: Non-Alcoholic Steatohepatitis; Bariatric Surgery; Gut Microbiota; Gut-Liver Axis; Metabolomics; Metagenomics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and portal vein (during operation) samples will be collected in this study. Plasma for biochemistry and metabolomics measurement, Buffy coat for NAFLD-susceptible single nucleotide polymorphism (SNP) detection (i.e. PNPLA3, TM6SF2...etc), peripheral blood mononuclear cell (PBMC) for flow cytometry, urine samples for lactulose/mannitol measurement (gut permeability test), fecal samples for metagenomics and metabolomics studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obese patients tissue proved NASH: age >20，morbid obesity who will receive bariatric surgery, tissue proved NASH
- Obese patients tissue proved NAFL: age >20，morbid obesity who will receive bariatric surgery, tissue proved NAFL
- NASH (before bariatric surgery): age >20，morbid obesity receiving bariatric surgery and was proved NASH histologically. Data collected before bariatric surgery.
  Interventions: Procedure: Bariatric surgery
- NASH (after bariatric surgery): age >20，morbid obesity receiving bariatric surgery and was proved NASH histologically. Data collected after bariatric surgery.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery
  Other Names: Liver biopsy; Portal vein sampling
  Groups: NASH (after bariatric surgery); NASH (before bariatric surgery)

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most common chronic liver disease. Non-alcoholic steatohepatitis (NASH) is an aggressive form of NAFLD with remarkable inflammatory features which may cause advanced fibrosis and liver cancer. So far there is no FDA-approved drug for treating NASH. A 10% weight loss by life style modification is a standard recommendation to treat NASH which achieves only 10-20% success rate in clinical practice. Thus, the development of therapeutics to prevent and treat NASH is certainly an unmet need. For now, the mechanism of how simple steatosis progresses to NASH remains unclear and accumulating evidences suggest the role of gut microbiota may be essential. Studies have also noted the bariatric surgery effectively improve diabetes and NASH with significant alterations in the composition and function of gut microbiome. In this study, the investigators aim to investigate the role of gut microbiota in the pathophysiology of NASH by comparing NAFLD severity, gut microbiome, metabolomics, immune profiles among patients before and after the bariatric surgery. With these efforts, the investigators wish to decipher the mechanism of how bariatric surgery may improve NASH through changing the gut microbiota and find out microbe-associated molecular signatures between NASH and NAFLD through this study.

DETAILED DESCRIPTION:
The investigators anticipate to recruit 140 morbidly obese patients who will receive bariatric surgery including 100 patients receiving sleeve gastrectomy (SG) and 40 receiving gastric bypass surgery (GB). Liver biopsy will be performed during the operation to confirm the histological scores of NAFLD severity. The investigators expect to have 50% NASH and 50% NAFL patients from these morbidly obese patients based on previous domestic data. (i.e. 50 patients receiving SG to have NASH and 50 patients receiving SG to have NAFL; 20 patients receiving GB to have NASH and 20 patients receiving GB to have NAFL.) In this study, the investigators have two study objectives which are as follows.

1. The first objective is to discover potential mechanisms among gut-liver axis for preventing or promoting NAFL to NASH by comparing (1) fecal microbiome composition and metabolomics, (2) peripheral blood biochemistry, metabolomics, immune cell phenotypes, and cytokines (3) portal vein biochemistry, metabolomics, immune cell phenotypes, and cytokines (4) Liver metabolomics and RNA-seq (5) gut permeability test (lactulose/mannitol challenge) (6) host genetic susceptibility for NAFLD (PNPLA3 and TM6SF2) between the tissue-proved NASH and NAFL patients in this study with a cross-sectional comparison.
2. The second objective is to longitudinally investigate the potential mechanisms of bariatric surgery for improving NASH via a gut-microbiota dependent pathway. Clinical and experimental data before (baseline) and after (1st, 3rd, 6th months) bariatric surgery will be collected which include (1) non-invasive evaluation of NAFLD severity (Fibroscan, MRI-PDFF (proton density fat fraction) and MRE), (2) blood biochemistry, metabolomics, immune cell phenotypes, and cytokines (3) fecal microbiome and metabolomics (4) gut permeability test (5) liver biopsy histology (if available)

ELIGIBILITY:
Inclusion Criteria:

Age >20，morbidly obese patients who will receive bariatric surgery.

Exclusion Criteria:

* Average daily alcohol intake >20 grams,
* Hepatitis B carriers, Hepatitis C carriers,
* people with liver disease caused by other causes
* liver cirrhosis,
* diseases related to abnormal blood coagulation,
* inflammatory bowel disease,
* routine use of steroids or immunity Inhibitors and other immunomodulatory drugs
* ursodeoxycholic and other drugs that affect bile acid metabolism
* those who have used antibiotics or probiotics within one month

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients who planned to receive bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of NAFLD severity score (histology) from baseline to the 6th month | Baseline and 6 months after bariatric surgery
  Liver biopsy will be performed before and after surgery (if available) to acquire histology evaluation
Change of NAFLD severity measured by Fibroscan from baseline to the 6th month | Baseline and 6 months after bariatric surgery
  Fibroscan (CAP and kPa)
Change of NAFLD severity measured by MRI proton density fat fraction from baseline to the | Baseline and 6 months after bariatric surgery
  MRI proton density fat fraction (%)
Change of NAFLD severity measured by magnetic resonance elastography from baseline to the | Baseline and 6 months after bariatric surgery
  magnetic resonance elastography (kPa)

SECONDARY OUTCOMES:
Change of gut microbiome profiles | Baseline, 1st month, 3rd month and 6th month after surgery
  fecal 16S ribosomal RNA sequencing and shotgun metagenome sequencing
Change of body fluid metabolomic profiles | Baseline, 1st month, 3rd month and 6th month after surgery
  Metabolites in blood fluids measured by liquid chromatography mass spectrometry
Change of Immune profiles | Baseline, 1st month, 3rd month and 6th month after surgery
  Immune cell phenotype patterns in body fluids measured by flow cytometry
Change of gut permeability test | Baseline and 6 months after bariatric surgery
  Lactulose/Mannitol challenge test
Change of gene expression profiles of liver tissue | Baseline and 6 months after bariatric surgery (if available)
  gene expression measured by RNA-seq
Change of metabolomic profiles of liver tissue | Baseline and 6 months after bariatric surgery (if available)
  Metabolites in liver tissue measured by liquid chromatography mass

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No